CLINICAL TRIAL: NCT04672733
Title: Hizentra® in Inflammatory Neuropathies - pHeNIx Study
Acronym: pHeNIx
Status: Recruiting | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: pHeNIx study; 2019-A01803-54 (Other: ANSM)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: CIDP; IgPro20; Hizentra; Subcutaneous Immunoglobulins
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Hizentra

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Hizentra — Solution for injection for subcutaneous use
  Other Names: IgPro20

SUMMARY:
The pHeNIx study, a national multicentre prospective non-interventional study, should help to describe the conditions of use for Hizentra® and the methods for switching from the IV to SC route in everyday practice, together with the tolerability and efficacy of treatment, which is monitored using a patient application (PRO: Patient-Reported Outcomes).

DETAILED DESCRIPTION:
Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) is a neurological and rare type of autoimmune disorder. Intravenous immunoglobulin (IVIg) is the first-line treatment for CIDP which has been proven to be effective. For several years, published cases have suggested that the Sub-Cutaneous Ig (SCIg) may be an alternative treatment to IVIg in the treatment of CIDP. Compared to IVIg treatment, the SCIg can achieve more stable plasma IgG concentrations, suggesting a potential reduction in the dose exhaustion effect at the end of the cycle, but also fewer systemic effects. SC administration also enables more straightforward treatment to be given for ambulatory patients.

Based on the PATH study (NCT01545076), a double blind placebo-controlled, randomised, prospective, international multicentre phase III study, Hizentra® obtained an extension of its marketing authorization for the CIDP indication as maintenance treatment after stabilisation with IVIg.

However, in the "real-life" situation, the literature is still based at present on small series of patient or short-term follow-up periods.

However, the methods for switching from the IV to the SC route and the characteristics of patients receiving this treatment are not known. In addition, SCIg administration remote from a specialist centre without assistance from a health professional no longer enables a more regular assessment of the patient in terms of tolerability and efficacy.

The pHeNIx study, a national multicentre prospective non-interventional study, should help to describe the conditions of use for Hizentra® and the methods for switching from the IV to SC route in everyday practice, together with the tolerability and efficacy of treatment, which is monitored using a patient application (PRO: Patient-Reported Outcomes). The study duration is estimated to be 36 months in view of: a 24-month inclusion period and a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (aged ≥18 years)
* Patients suffering from CIDP according to EAN/PNS 2021 criteria
* Planned switch from IVIg to Hizentra®
* Patient treated with at least 3 courses of IV immunoglobulin and deemed by the investigator to be dependent on immunoglobulins
* Patient deemed to be stable, with no change in their treatment for the disease during the 3 months prior to inclusion
* Patients who have a smartphone, a tablet or a computer
* Patients who have been informed verbally and in writing of the purposes of the study

Exclusion Criteria:

* Concomitant participation in an interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French cohort of patients with CIDP
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Length of time of Continuation of treatment | up to 12 months
  Non-continuation is defined by:
  * an increase in the INCAT score of over one point measured in a consultation despite a bolus dose of IVIg and/or after increasing the dose of Hizentra®
  * stopping treatment with Hizentra®

SECONDARY OUTCOMES:
The time between the last dose of IVIg and starting Hizentra® | At Baseline
The total dose of the last course of IVIg | At Baseline
The interval between courses of IVIg | At Baseline
The total dose of the first course of Hizentra | At Baseline
The number of days of the first course of Hizentra | At Baseline
Number of Self-administrations or administrations by a state-registered nurse | Up to 12 months
The daily dose of Hizentra | Up to 12 months
The daily volume of Hizentra | Up to 12 months
Duration of the infusion | Up to 12 months
Number of infusion sites | Up to 12 months
Number of Patients completing the Patient Reported Outcome (PRO) tests at home | Up to 12 months
Rasch-built Overall Disability Scale (RODS) incapacity scale score by patient | Up to 12 months
10-metre walking test score by patient | Up to 12 months
Rasch-built Overall Disability Scale (RODS) incapacity scale score by doctor | Up to 12 months
10-metre walking test score by doctor | Up to 12 months
Time since the diagnosis of CIDP | At baseline
EuroQol-5D (EQ-5D) quality of life score | Up to 12 months
Pictorial Representation of Illness and Self Measure (PRISM) score | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring SA
Locations (27):
- France (27):
  - CHU Amiens Picardie 1, Amiens
  - CHU Angers, Angers
  - Hôpital privé de La Casamance, Aubagne
  - CH Bayonne, Bayonne
  - Hôpital Pellegrin, Bordeaux
  - CHRU Brest, Brest
  - Hôpital Henri Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH Libourne, Libourne
  - Hôpital Roger Salengro, CHU Lille, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital Pierre Wertheimer,HCL, Lyon
  - Hôpital de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Lariboisière, Paris
  - La Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - Centre hospitalier privé Saint Grégoire, Rennes
  - Hôpital Charles Nicolle, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHR Tours, Tours
  - CH de Valence, Valence